CLINICAL TRIAL: NCT07264816
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of BL-M07D1 in Combination With Pembrolizumab in Patients With Unresectable Locally Advanced or Metastatic HER2-Overexpressing Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of BL-M07D1 in Combination With Pembrolizumab in Patients With Unresectable Locally Advanced or Metastatic HER2-Overexpressing Non-Squamous NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M07D1-207
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-M07D1+pembrolizumab (Experimental): Participants received BL-M07D1+pembrolizumab in the first cycle (3 weeks). Participants who had a clinical benefit could receive additional cycles of additional treatment. Administration will be discontinued because of disease progression or intolerable toxicity or for other reasons.
  Interventions: Drug: BL-M07D1; Drug: Pembrolizumab

INTERVENTIONS:
Drug: BL-M07D1 — Administration by intravenous infusion for a cycle of 3 weeks.
Drug: Pembrolizumab — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This trial is a multicenter, open-label, Phase II clinical study to explore the efficacy and safety of BL-M07D1 in combination with pembrolizumab in patients with locally advanced or metastatic HER2-overexpressing non-squamous non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements;
2. No gender restrictions;
3. Age at the time of signing the informed consent form ≥18 years and ≤75 years;
4. Expected survival time ≥3 months;
5. Patients with locally advanced or metastatic non-squamous non-small cell lung cancer;
6. Confirmed known HER2 overexpression;
7. Agree to provide archived tumor tissue specimens from primary or metastatic lesions within the past 2 years;
8. Must have at least one measurable lesion meeting the RECIST v1.1 criteria;
9. ECOG performance status score of 0 or 1;
10. Toxicities from prior anti-tumor treatments have recovered to ≤ Grade 1 as defined by NCI-CTCAE v5.0;
11. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
12. Organ function levels must meet the requirements;
13. For premenopausal women with childbearing potential, a pregnancy test must be conducted within 7 days before starting treatment, serum pregnancy must be negative, and they must not be breastfeeding; all enrolled patients (regardless of gender) should take adequate and highly effective contraception throughout the treatment cycle and for 7 months after the end of treatment.

Exclusion Criteria:

1. Underwent surgical treatment, radical radiotherapy, immunotherapy, etc., within 4 weeks before the first dose or within 5 half-lives;
2. Pathology indicates non-small cell carcinoma containing small cell carcinoma components and sarcomatoid carcinoma;
3. Previously received HER2-targeted therapy or ADC drug treatment with camptothecin derivatives as toxins;
4. History of severe cardiovascular or cerebrovascular diseases within the past 6 months before screening;
5. Concurrent pulmonary disease leading to severe impairment of lung function;
6. QT interval prolongation, complete left bundle branch block, third-degree atrioventricular block, frequent and uncontrollable arrhythmias;
7. Diagnosed with other primary malignancies within 5 years before the first dose;
8. Poorly controlled hypertension;
9. History of non-infectious ILD requiring steroid treatment, or currently suffering from ILD/interstitial pneumonia, etc.;
10. Patients with central nervous system metastases, carcinomatous meningitis, and/or spinal cord compression;
11. Patients with a history of allergy to recombinant humanized antibodies or allergy to BL-M07D1, pembrolizumab, or any excipient components;
12. Required systemic corticosteroid or immunosuppressive therapy within 2 weeks before the study administration;
13. Patients with massive serous cavity effusion, symptomatic serous cavity effusion, or poorly controlled serous cavity effusion;
14. New deep vein thrombosis within 14 days, excluding patients with venous filters implanted;
15. Systemic severe infection within 4 weeks before screening;
16. Active autoimmune diseases and inflammatory diseases;
17. Human immunodeficiency virus antibody positivity, active hepatitis B virus infection, or hepatitis C virus infection;
18. History of allogeneic stem cell, bone marrow, or organ transplantation;
19. Presence of severe neurological or psychiatric disorders;
20. Presence of other severe physical or laboratory abnormalities, poor compliance, etc., which may increase the risk of participation in the study, interfere with study results, or patients deemed unsuitable for participation in the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Combined optimal dosage | Up to approximately 24 months
  The combined optimal dosage will be investigated.
Combination method | Up to approximately 24 months
  The combination method will be investigated.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-M07D1 to the first date of either disease progression or death, whichever occurs first.
Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of BL-M07D1 will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of BL-M07D1 will be investigated.
Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of BL-M07D1 prior to the next dose will be administered.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-BL-M07D1 antibody (ADA) will be investigated.
Drug-drug interactions (DDI) | Up to approximately 24 months
  Drug-drug interactions (DDI) will be investigated.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M07D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M07D1.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China